CLINICAL TRIAL: NCT00433693
Title: Correction Study of Intravenous Injections of R744 to Hemodialysis Patients ( Phase Ⅲ Study ).
Brief Title: Correction Study of R744 in Renal Anemia Patients on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JH20562
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Hemodialysis Patients
MeSH Terms: interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: R744

INTERVENTIONS:
Drug: R744 — 50μg(i.v.)/2 week until Hb concentration reaches to 11.0g/dL or above, then 25~300μg(i.v.)/4 week
  Other Names: methoxy polyethylene glycol-epoetin beta

SUMMARY:
This study will assess the efficacy and safety of intravenous R744 in renal anemia patients on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been receiving hemodialysis more than 1 time a week
* Patients aged ≥ 20 years at the time of obtaining consent
* After starting of hemodialysis, patients who have not received rHuEPO preparation
* After starting of hemodialysis, patients whose value of Hb concentrations determined before the first hemodialysis during the last week prior to the registration has been < 10.0 g/dL

Exclusion Criteria:

* Patients with hardly controllable hypertension (patients whose diastolic blood pressure has been ≥ 100 mmHg on more than 1/3 of the determining occasions after starting of hemodialysis during the last week before registration)
* Patients with congestive cardiac failure (≥ Class III in NYHA cardiac function classification)
* Female patients who are pregnant, lactating, possibly pregnant or not willing to take a contraceptive measure during the period from the day of starting the treatment with the study drug to 90 days after the day of the last dose of the study drug
* Patients with complication of myocardial infarction, pulmonary infarction or cerebral infarction (excluding asymptomatic cerebral infarction)
* Patients confirmed to have serious allergy or serious drug allergy (shock, anaphylactoid symptom)
* Patients hypersensitive to a rHuEPO preparation
* Patients with malignant tumor (including hemic malignant tumor), severe infection, systemic hemic disease (osteomyelodysplasia syndrome, hemoglobinopathy, etc.), hemolytic anemia or apparent hemorrhagic lesion such as digestive tract hemorrhage
* Patients who have received an anabolic hormone preparation, testosterone enanthate or mepitiostane within 12 weeks before registration
* Patients who have received another investigational drug within 12 weeks before registration
* Patients who have received R744 before registration
* Patients whose AST(GOT) value ≥ 100 IU/L or ALT(GPT) value ≥ 100 IU/L before registration
* Patients who have received erythrocyte transfusion within 16 weeks before registration
* Patients for whom a surgical operation involved with heavy bleeding is planned during the study period
* In addition, patients who are judged as ineligible to participate in this study by the investigator or sub-investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The ratio of patients whose Hb concentration reach ≥ 10.0g/dL and increasing amount of Hb concentration reach ≥ 1.0g/dL | 26 weeks

SECONDARY OUTCOMES:
Time required for reaching Hb concentration of ≥ 10.0 g/dL and reaching increasing amount of Hb concentration ≥ 1.0g/dL | 26 weeks
Regression line of Hb concentration per week | 26 weeks
Achievement rate of Hb concentration of ≥ 11.0 g/dL | 26 weeks
Transition of Hb concentration | 26 weeks
dose transition of study drug | 26 weeks
Variation of QOL | 26 weeks
Adverse events | 26 weeks
Laboratory measurements | 26 weeks
Vital signs, standard 12-lead ECG | 26 weeks
Anti-R744 antibody titer | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Takanori Baba, Study Chair — Clinical Research Department 2
Locations (6):
- Japan (6):
  - Chugoku/Shikoku region, Chugoku/Shikoku
  - Chubu region, Chūbu
  - Hokkaido/Tohoku region, Hokkaido/Tohoku
  - Kanto/Koshinetsu region, Kanto/Koshinetsu
  - Kinki/Hokuriku region, Kinki/Hokuriku
  - Kyusyu region, Kyusyu